CLINICAL TRIAL: NCT06398015
Title: Open Surgical Reconstruction Versus Open Sham Surgery in the Treatment of Hip Abductor Tendon Tears; A Double Blinded, Randomized Controlled Trial
Brief Title: Hip Abductor Tendon Repair Versus Sham Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horsens Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Jeppe Lange, MD, PhD, Horsens Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-16-02-128-24
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Rupture of Hip Abductor Tendon (Disorder)
Keywords: orthopedics; hip injuries; rehabilitation; sham surgery; lateral hip pain; hip abductor tendon tear
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients are allocated when in full general anesthesia. Treatment allocation will be blinded in the electronic patient journal, as the surgeon will insert a general description of the surgery. Unblinding at 6 months at the final consultation with the orthopedic surgeon. At the day of the unblinding the patient will be tested in the Department of Physio- and Occupational Therapy before the consultation with the orthopedic surgeon.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rHat-group (Experimental): Surgical reconstruction of hip abductor tendon tear
  Interventions: Procedure: Surgical reconstruction of hip abductor tendon tear
- SHAM-group (Sham Comparator): Sham surgery of hip abductor tendon tear
  Interventions: Procedure: Sham surgery of hip abductor tendon tear

INTERVENTIONS:
Procedure: Surgical reconstruction of hip abductor tendon tear — If the patient is allocated to surgical reconstruction, the incision from the sham surgery is continued into the iliotibial band (ITB) and down to the hip abductor tendon complex/greater trochanter. A standardized reconstruction of the HAT with bone anchors is then performed.
  This standardized procedure has been used by the surgeons for the last 6 years. The ITB is then closed with looped suture, the subcutaneous tissue sutured with standard resorbable single sutures, the skin stapled and a standard wound dressing is applied.
  Arms: rHat-group
Procedure: Sham surgery of hip abductor tendon tear — If the patient is allocated to sham surgery, the incision will only include the skin and subcutaneous tissue. Subsequently, the subcutaneous tissue will be sutured with standard resorbable single sutures, the skin stapled and a standard wound dressing applied. The patient will be kept in general anesthesia for 10 minutes after the procedure is finalized to mimic a true intervention (to hinder staff or relatives to comment on the duration of the procedure). The normal standard procedure takes approximately 40 minutes.
  Arms: SHAM-group

SUMMARY:
This study will examine the effectiveness of open surgical reconstruction in the treatment of patients with hip abductor tendon tears. Patients will be randomly allocated to either the open surgical reconstruction or to a open surgical sham procedure. The primary outcome is patient reported pain measured by the revised Copenhagen Hip And Groin Outcome Score (HAGOS), which will be conducted pre-surgery and at three and six months post-surgery. The six-month follow-up is the primary endpoint.

DETAILED DESCRIPTION:
This is a study protocol for a Good Clinical Practice-monitored, double-blinded, randomized, controlled superiority trial with two groups, where the primary endpoint is differences in changes in lateral hip pain 6 months post-surgery. If included in the study, patients will be randomly allocated to one of the two arms:

1. Open surgical reconstruction of the hip abductor tear (rHAT-group)
2. Sham surgery (SHAM-group)

Patients will be allocated with a 1:1 ratio using permuted blocks with random varying sizes of 4, 6, and 8. An interim analysis will be performed when 8 patients in each group have completed the primary outcome assessment at 6 months.

Post-surgery, the patients in both groups will be guided and instructed in exercises according to their pain levels and functional capacity by an experienced physiotherapist blinded to the allocation. The first 6 post-surgery weeks, rehabilitation is home-based. After the 6-week follow-up, the patients will be referred to further rehabilitation in their home municipality (current standard practice).

The patients will be assessed pre-surgery, at 3 months post-surgery, and at the final follow-up at 6 months post-surgery. A physiotherapist blinded to the allocation will test the patients at the abovementioned timepoints.

In the trial paper all outcomes conducted will be published. That is, the primary outcome and the following secondary outcomes: The remaining five subscales of the revised HAGOS questionnaire (symptoms, function in daily living, function in sport and recreation, participation in physical activity, quality of life), Oxford Hip Score (OHS), European Questionnaire-5 Dimension (EQ-5D-5L and EQ-VAS), Global Rating of Change (GroC), Lateral hip pain on a numerical rating scale (NRS), The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G), isometric hip abduction muscle strength, functional capacity by a 30 second Chair Stand Test (30s-CST).

The primary aim is to evaluate between-group changes on hip pain based on the subscale "pain" from the patient-reported outcome measure the revised Copenhagen Hip And Groin Outcome Score (HAGOS) from pre-surgery to 6 months post-surgery.

Primarily The primary hypothesis: The score in the subscale "pain" on the revised HAGOS will increase more in the intervention group compared to the control group, 6 months post-surgery.

A full study protocol will be published and made available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an MRI verified hip abductor tendon pathology
* Age 30 years or above
* Lateral hip pain for more than 12 months
* Ability to understand written and verbal Danish

Exclusion Criteria:

* Previous hip joint replacement, pelvic osteomies, hip abductor tendon surgery, femoral nailing or iliotibial band surgery
* Pregnancy
* Osteoarthritis of the hip joint on the affected side (Kellgren Lawrence grade +2)
* Rheumatoid disorders
* Inability to attend planned follow-up visits
* Having an ongoing occupational injury insurance case
* Expected lack of compliance due to cognitive issues, alcohol, or drug abuse

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Differences in changes in patient-reported pain measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The subscale "pain" on HAGOS measures the patients perception of hip and/or groin pain. It consist of ten items. A score from 0 to 100 is calculated, where a higher score is indicating lower pain.

SECONDARY OUTCOMES:
Differences in changes in patient-reported symptoms measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The subscale "symptoms" on HAGOS measures the patients perception of hip and/or groin pain. It consist of seven items. A score from 0 to 100 is calculated, where a higher score is indicating lower symptoms.
Differences in changes in patient-reported physical function in daily living (ADL) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The subscale "ADL" on HAGOS measures the patients perception of hip and/or groin pain. It consist of five items. A score from 0 to 100 is calculated, where a higher score is indicating higher function.
Differences in changes in patient-reported physical function in sport and recreational activities (sport/recreation) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The subscale "sport/recreation" on HAGOS measures the patients perception of hip and/or groin pain. It consist of eight items. A score from 0 to 100 is calculated, where a higher score is indicating higher function.
Differences in changes in patient-reported participation in physical activities (PA) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The subscale "PA" on HAGOS measures the patients perception of hip and/or groin pain. It consist of two items. A score from 0 to 100 is calculated, where a higher score is indicating higher ability to participate in physical activity.
Differences in changes in patient-reported quality of life (QOL) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The subscale "QOL" on HAGOS measures the patients perception of hip and/or groin pain. It consist of five items. A score from 0 to 100 is calculated, where a higher score is indicating higher quality of life.
Differences in changes in the patient-reported outcome measure Oxford Hip Score (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  Oxford Hip Score (OHS), which consists of 12items. OHS is developed and validated for patients undergoing total hip replacements to access pain and function. It is a composite score ranging from 0 (worst) to 48 (best).
Differences in changes in the patient-reported outcome measure EQ-5D-5L (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  European Questionnaire-5 Dimensions (EQ-5D-5L and EQ-VAS) consists of five items and a visual analogue score (VAS), a vertical line on which the patients score their perception of their overall health from 0 to 100 (worst to best)
Global Rating of Change (GRoC) | The outcome is conducted at 3- and 6-months post-surgery follow-up.
  GRoC consists of a 11-point scale, where the patient rates the perceived overall change of the hip condition from "very much better" to "very much worse" . Responses on GRoC will be considered successful if patients scored "moderately better" to "very much better". Global improvement will be measured as the percentage of successful reports.
Differences in changes in lateral hip pain on a numerical pain rating scale (NRS) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  Participants rate their pain on a scale from 0 (no pain) to 10 (worst imaginable). Participants will rate their average pain for the past 14 days during rest and activity.
Differences in changes in the patient-reported outcome measure The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) is validated for patients with gluteal tendinopathy and measures the severity of disability related to the condition. VISA-G consist of eight items and appraise the pain in relation to gluteal tendinopathy by a score from 0-100, where a higher score will indicate lower pain and less disability.
Differences in changes of maximal isometric hip abduction muscle strength (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  Maximal isometric hip abduction strength test measures the maximal voluntary isometric contraction in supine position. The strength will be measured using a fixed dynamometer. Strength will be conducted in Newton, but will be normalised according to the lever arm and body weight, and will be reported as Nm/kg bodyweight.
Differences in changes of the number of repetitions of a 30 second sit to stand test (continuous data) | From baseline to 6-months post-surgery follow-up. The outcome is also conducted at 3-months post-surgery follow-up.
  Number of repetitions (sits to stand) performed during 30 seconds on a chair with a seat height of 46 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Høgsholt, PT, PhD.st., Principal Investigator — Horsens Regional Hospital; Aarhus University; Jeppe Lange, MD, PhD, Study Director — Horsens Regional Hospital; Aarhus University; Signe Kierkegaard-Brøchner, PhD, Study Chair — Regionshospitalet Horsens; Kristian Thorborg, PhD, Study Chair — Copenhagen University Hospital, Hvidovre; Marie Bagger Bohn, MD, PhD, Study Chair — Regionshospitalet Horsens
Locations (1):
- Horsens Regional Hospital, Horsens, Denmark

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared: All quantitative individual participant data collected during the trial, after deidentification, and according to current Danish Data Protection Regulation and GDPR.
  With whom will data be shared: Researchers who provide a methodologically sound proposal.
  For what types of analyses: To achieve aims in the approved proposal. The abovementioned is based on Data Sharing Statements for Clinical Trial: A Requirement of the ICMJE located at: https://www.icmje.org/news-and-editorials/data_sharing_june_2017.pdf
Supporting Information: Study Protocol
Time Frame: Immediately following publication and ending 5 years following primary article publication.
Access Criteria: Proposals should be directed to mathhg@rm.dk. To gain access, data requestors will need to sign a data access agreement.